CLINICAL TRIAL: NCT00120926
Title: Randomized Control Trial Evaluating the Effect of Two Different Doses of Amino Acids on Growth and Serum Amino Acids in Premature Neonates Admitted to the NICU
Brief Title: Dose Comparison of Amino Acids on Growth in Premature Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pediatrix (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDX05-001
Record Dates: First submitted 2005-07-11; First posted 2005-07-19 (Estimated); Last update posted 2006-09-28 (Estimated); Status verified 2006-09

CONDITIONS: Malnutrition
Keywords: Premature neonate; Parenteral nutrition; Growth; Amino Acids; Nutrition
MeSH Terms: conditions — Malnutrition; Premature Birth; Hyperphagia | interventions — Parenteral Nutrition

INTERVENTIONS:
Drug: Parenteral Nutrition

SUMMARY:
Malnutrition is a common problem in the neonatal intensive care unit. Recent studies indicate that prematurely born neonates commonly develop a severe nutritional deficit during the first weeks after birth, referred to as extrauterine growth restriction. Despite an increase in growth during the second month of hospitalization, many neonates are ultimately discharged home having grown inadequately. The early nutritional deficit affects weight gain as well as growth in length and head circumference.

Growth measurements such as weight, length, and head circumference, however, are macroscopic measures of nutritional status and underestimate the physiologic consequences of prolonged nutritional deprivation. Energy and micronutrient deficiencies alter growth at a cellular and tissue level before macroscopic measures are altered. In the brain, for instance, energy is required for cell division and neuronal growth, glial cell function, and myelination. Energy deprivation may consequently alter neuronal function and growth, resulting in adverse neurodevelopmental outcomes.

Immunocompetence also appears to be sensitive to the untoward effects of energy and nutritional deficiency. Malnourished neonates often exhibit immune deficiencies related to inadequate protein intake that compound an already immature immune system. Such immunodeficiency results in susceptibility to infectious agents that creates substantial morbidity and mortality to the course of intensive care for premature infants.

A recent study suggests that postnatal malnutrition and growth restriction are inevitable if current recommended dietary intakes are followed. Multicenter studies show that variation in dietary intake accounts for 45% of the variation in growth. Hence, efforts have focused on determining whether nutritional deficiency and the observed growth restriction of premature infants can be prevented through the use of more optimal nutritional intake. In addition, inadequate protein support may be a primary cause for growth failure.

Based on animal studies showing high in utero amino acid flux observed during the latter phase of gestation, Thureen et al have suggested the use of higher doses of amino acid supplementation in order to minimize growth restriction and improve outcomes of premature infants. However there are no large human trials that demonstrate that this approach promotes better growth or that it is safe. While small doses of amino acids may be inadequate to promote normal growth, high doses may lead to elevated serum amino acid levels and increase the occurrence of toxicity. Through the implementation of a multicenter, randomized trial and tandem mass spectrometry, the investigators propose to evaluate the effects of two distinct strategies of amino acid supplementation on serum amino acid profiles and growth of premature infants during the first 28 days of life.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of informed consent
* Inborn
* Gestational age between 23 weeks and 0/7 days and 29 weeks and 6/7 days
* If subject is transferred to another hospital, the ability to obtain follow-up data on outcomes
* No major anomalies
* Ability to begin parenteral nutrition within the first 48 hours after birth

Exclusion Criteria:

* Outborn
* Gestational age < 23 weeks or >= 30 weeks
* Any major congenital anomalies

Ages: 0 Years to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2005-08; Study Completion 2006-06

PRIMARY OUTCOMES:
The primary outcome is growth velocity for first 28 days of life calculated as: weight gain, head circumference, length

SECONDARY OUTCOMES:
Secondary outcomes include serum amino acid profiles measured on: day 7 of life, day 28 of life

CONTACTS AND LOCATIONS:
Overall Officials: Reese Clark, MD, Principal Investigator — Pediatrix Medical Group, Inc.
Locations (1):
- McLeod Regional Medical Center, Florence, South Carolina, United States

REFERENCES:
- [Background] Thureen PJ, Melara D, Fennessey PV, Hay WW Jr. Effect of low versus high intravenous amino acid intake on very low birth weight infants in the early neonatal period. Pediatr Res. 2003 Jan;53(1):24-32. doi: 10.1203/00006450-200301000-00008. PMID 12508078
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765
- [Derived] Kelleher AS, Clark RH, Steinbach M, Chace DH, Spitzer AR; Pediatrix Amino-Acid Study Group. The influence of amino-acid supplementation, gestational age and time on thyroxine levels in premature neonates. J Perinatol. 2008 Apr;28(4):270-4. doi: 10.1038/jp.2008.5. Epub 2008 Feb 21. PMID 18288119
- [Derived] Steinbach M, Clark RH, Kelleher AS, Flores C, White R, Chace DH, Spitzer AR; Pediatrix Amino-Acid Study Group. Demographic and nutritional factors associated with prolonged cholestatic jaundice in the premature infant. J Perinatol. 2008 Feb;28(2):129-35. doi: 10.1038/sj.jp.7211889. Epub 2007 Dec 6. PMID 18059467
- [Derived] Clark RH, Chace DH, Spitzer AR; Pediatrix Amino Acid Study Group. Effects of two different doses of amino acid supplementation on growth and blood amino acid levels in premature neonates admitted to the neonatal intensive care unit: a randomized, controlled trial. Pediatrics. 2007 Dec;120(6):1286-96. doi: 10.1542/peds.2007-0545. PMID 18055678
- See also: Related Info — http://www.pediatrix.com